CLINICAL TRIAL: NCT03334032
Title: Incomplete Total Body Protein Recovery in Adolescent Patients With Anorexia Nervosa
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: University of Sydney (Other)
Responsible Party: Principal Investigator, Dr. Verena Haas, Principle Investigator, Clinical Researcher, Charite University, Berlin, Germany
Other Study IDs: TBN in AN
Record Dates: First submitted 2017-10-29; First posted 2017-11-07 (Actual); Last update posted 2017-11-07 (Actual); Status verified 2017-11

CONDITIONS: Anorexia Nervosa
Keywords: Body composition; Total body protein; nutritional recovery; Exercise status; In-vivo neutron activation analysis; Protein depletion
MeSH Terms: conditions — Anorexia Nervosa | interventions — Hospitalization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Inpatient treatment for Anorexia nervosa: Adolescents with anorexia nervosa assessed
  1. at baseline: on admission to inpatient treatment
  2. at follow-up: 6 months after admission on outpatient basis
  Interventions: Other: Inpatient treatment for Anorexia nervosa
- Controls: Adolescent healthy and normal weight controls (matched for gender and age), assessed at one point of time

INTERVENTIONS:
Other: Inpatient treatment for Anorexia nervosa — Nutritional rehabilitation in a clinic with specialized eating disorder service
  Groups: Inpatient treatment for Anorexia nervosa

SUMMARY:
The study aimed to assess protein accretion during weight gain in adolescent patients with Anorexia nervosa

DETAILED DESCRIPTION:
Background: Bone health and growth during adolescence require adequate Total Body Protein (TBPr). Re-nutrition for patients with anorexia nervosa (AN) should aim to normalize body composition, i.e. recovery of fat mass and TBPr.

Objective: The study intended to analyze predictors of protein status, including exercise status, in adolescents with AN, and to investigate whether weight gain would replete body protein deficits.

Methods: The investigators assessed TBPr in a longitudinal, observational study as height-adjusted nitrogen index (NI) using in-vivo neutron activation analysis in adolescents with AN at the commencement of refeeding (T0), as well as seven months thereafter (T1), and in age-matched normal weight controls. Lean tissue and fat mass were assessed with Dual-Energy X-Ray Absorptiometry (DXA). BMI, BMI-SDS and lean tissue mass were tested as predictors of protein status using Receiver Operating Characteristic (ROC) analysis.

ELIGIBILITY:
Patient Inclusion Criteria:

* diagnosis of anorexia nervosa (DSM-IV)
* aged 12 - 19 years
* female gender

Patient Exclusion Criteria:

- existence of a further disease with effect on body composition

Controls:

* no known disease
* normal weight

Ages: 12 Years to 19 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: At baseline assessment, ten patients had primary amenorrhea and 87 girls secondary amenorrhea. Six girls were not amenorrhoeic but were taking oral contraceptives or had lost more than 20% of their weight and fulfilled the remaining diagnostic criteria for AN. The mean duration of the eating disorder at the time of testing was 15 ± 12 months, ranging from 3 to 60 months and estimated premorbid BMI of the AN patients was 20.4 ± 2.9 (13.5 - 28.7 kg/m2; data available for 98 patients). Before admission, the patients (n = 97) had lost 15 ± 7 (2 - 36) kg. The mean weight on hospital admission (data available for 88 patients; 10 patients were outpatients; missing data, n = 5) was 41.1 ± 6.1 kg.
Sampling Method: Non-Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2004-07 (Actual); Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change in Total Body protein | Between baseline (inpatient admission) and at 7 months follow-up
  Change in Total Body protein

SECONDARY OUTCOMES:
Change in body weight | Between baseline (inpatient admission) and at 7 months follow-up
  Change in: body weight (kg)
Change in Body Mass Index | Between baseline (inpatient admission) and at 7 months follow-up
  Change in Body Mass Index (BMI; kg/m2)
Change in body fat mass | Between baseline (inpatient admission) and at 7 months follow-up
  Change in body fat mass (kg)
Change in body lean tissue mass | Between baseline (inpatient admission) and at 7 months follow-up
  Change in body lean tissue mass (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Michael R Kohn, Prof., Principal Investigator — University of Sydney

IPD SHARING:
Plan to Share IPD: Undecided